CLINICAL TRIAL: NCT04088864
Title: Phase Ib Clinical Trial of Autologous CD22 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory B Cell Malignancies
Brief Title: CD22-CAR T Cells in Children and Young Adults With B Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-50878; CCT6003 (Other: OnCore); IRB-50878 (Other: Stanford IRB); NCI-2019-07285 (Other: NCI Trial Identifier)
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: B Cell Lymphoma; Acute Lymphoblastic Leukemia, Pediatric; Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- R/R B-ALL (Experimental): Subjects will receive a conditioning lymphodepletion chemotherapy regimen of fludarabine and cyclophosphamide followed by infusion of CD22 CAR T cells on Day0.
  Lymphodepletion:
  * Fludarabine 25 mg/m2 per day IV for days 4, 3, -2
  * Cyclophosphamide 900 mg/m2 per day IV on day -2
  Autologous CD22 CAR T cells will be administered intravenously at Dose level 1 (1 x 10^6 transduced T cells/kg (± 20%)).
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Autologous CD22 CAR T
- Lymphoma (Experimental): Subjects will receive a conditioning lymphodepletion chemotherapy regimen of fludarabine and cyclophosphamide followed by infusion of CD22 CAR T cells on Day0.
  Lymphodepletion:
  * Fludarabine 25 mg/m2 per day IV for days 4, 3, -2
  * Cyclophosphamide 900 mg/m2 per day IV on day -2
  Autologous CD22 CAR T cells will be administered intravenously at Dose level 1 (1 x 10^6 transduced T cells/kg (± 20%)).
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Autologous CD22 CAR T

INTERVENTIONS:
Drug: Fludarabine — Fludarabine is a purine antagonist antimetabolite
Drug: Cyclophosphamide — Cyclophosphamide is a nitrogen mustard derivative alkylating agent
Drug: Autologous CD22 CAR T — Autologous T cells transduced with lentiviral vector (m971BBZ) Chimeric Antigen Receptor (CD22 CAR)

SUMMARY:
The primary purpose of this study is to test whether CD22-CAR T cells can be successfully made from immune cells collected from pediatric and young adult subjects with relapsed/refractory B-cell malignancies (leukemia and lymphoma). Another purpose of this study is to test the safety and cancer killing ability of a cell therapy against a new cancer target (CD22).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* Determine the feasibility of manufacturing CD22 CAR T cells for administration to children and young adults with relapsed/refractory (R/R) CD22 expressing B-cell ALL or lymphoma using the Miltenyi CliniMACS Prodigy system.
* Determine the safety of an established dose of CD22-CAR T cells in children and young adults with R/R CD22 expressing B-cell malignancies.

SECONDARY OBJECTIVE:

- Assess the clinical activity of CD22-CAR T cells in children and young adults with R/R CD22 expressing B-cell malignancies, including overall survival (OS) and progression free survival (PFS).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Disease Status Disease Status of ALL

   * Must have chemotherapy refractory disease defined as progression or stable disease after two lines of therapies, or
   * Relapsed disease after achieving CR.
   * Subjects with persistent or relapsed minimal residual disease (MRD) (by flow cytometry, PCR, fluorescence in situ hybridization (FISH), or next generation sequencing (NGS) require verification of MRD on two occasions at least 2 weeks apart.
   * Subjects with Philadelphia Chromosome positive acute lymphoblastic leukemia (Ph+ALL) subjects are eligible if they progressed, had stable disease or relapsed after two lines of therapy, including tyrosine kinase inhibitors (TKIs).
   * Subjects with recurrence of isolated central nervous system CNS) relapse after achieving complete remission (CR).

   Disease Status of lymphoma
   * Histologically confirmed aggressive B cell NHL including the following types defined by WHO 2008:

     - DLBCL not otherwise specified; T cell/histiocyte rich large B cell lymphoma; DLBCL associated with chronic inflammation; Epstein Barr virus (EBV)+ DLBCL of the elderly; OR primary mediastinal (thymic) large B cell lymphoma transformation of follicular lymphoma, marginal zone lymphoma or chronic lymphocytic leukemia/small lymphocytic lymphoma to DLBCL will also be included
   * Subjects with DLBCL must have progressed, had SD, or recurred after initial treatment regimens that include an anthracycline and an anti CD20 monoclonal antibody. Subjects with transformed Follicular lymphoma(FL), marginal zone B-cell lymphoma (MZL), or chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) must have progressed, had SD, or recurred with transformed disease after initial treatment for DLBCL. Subjects who relapse ≥12 months after therapy should have progressed after autologous transplant or been ineligible for autologous transplant.
2. Measureable Disease

   * Subjects with ALL must have evaluable or measurable disease.
   * Subjects with lymphoma: Must have evaluable or measurable disease according to the revisedInternational Working. Group( IWG) Response Criteria for Malignant Lymphoma. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
3. CD22 expression

   • Subjects with ALL: CD22 positive expression on malignant cells is required and must be detected by immunohistochemistry or by flow cytometry. The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each subject.

   CD22 expression must be demonstrated subsequent to any anti-CD22 targeted therapy (e.g. Moxetumomab pasudotox or inotuzumab ozogamicin) in subjects with ALL

   • Subjects with lymphoma: must have archival tissue available for analysis of CD22 expression, or must be willing to undergo a biopsy of easily accessible disease.
4. Prior Bone Marrow-Stem Cell Transplant Subjects who have undergone autologous stem cell transplant (SCT) with disease progression or relapse following SCT are eligible. Subjects who have undergone allogeneic SCT will be eligible if, in addition to meeting other eligibility criteria, they are at least 100 days post transplant, they have no evidence of Graft versus host disease (GVHD) and have been without immunosuppressive agents for at least 30 days.
5. Prior Therapy Wash-out

   * At least 2 weeks or 5 half lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half lives.
   * Subjects with ALL may not have receive inotuzumab ozogamicin therapy within the past 4 months.

   Exceptions:
   * There is no time restriction with regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such;
   * Subjects receiving hydroxyurea may be enrolled provided there has been no increase in dose for at least 2 weeks prior to starting apheresis;
   * Subjects who are on standard ALL maintenance type chemotherapy (vincristine, 6- mercaptopurine or oral methotrexate) may be enrolled provided that chemotherapy is discontinued at least 1 week or 5 half-lives, whichever is shorter,prior to apheresis.
   * Subjects receiving steroid therapy at physiologic replacement doses (≤ 5 mg/day of prednisone or equivalent doses of other corticosteroids) only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis;
   * For radiation therapy: Radiation therapy must have been completed at least 3 weeks prior to enrollment, with the exception that there is no time restriction if the volume of bone marrow treated is less than 10% and also the subject has measurable/evaluable disease outside the radiation port or the site of radiation has documented progression.
6. Prior CAR Therapy Subjects who have undergone prior CAR therapy will be eligible if at least 30 days has elapsed prior to apheresis.
7. Toxicities from Prior Therapy Toxicities due to prior therapy must be stable (except for clinically non significant toxicities such as alopecia)
8. Age greater than or equal to 1 year and ≤ 30 years of age at time of enrollment. First 3 subjects treated at the dose level must be at least 16 years old (enrolled on either pediatric or adult protocol).
9. Performance Status:

   Subjects > 10 years of age: Karnofsky ≥ 70% OR Eastern cooperative oncology group (ECOG) performance status of 0 or 1; Subjects ≤ 10 years of age: Lansky scale ≥ 70%
10. Normal Organ and Marrow Function (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion)

    * Absolute neutrophil count (ANC) ≥ 750/uL*
    * Platelet count ≥ 50,000/uL*
    * Absolute lymphocyte count ≥ 150/uL*

    Adequate renal, hepatic, pulmonary and cardiac function defined as:
    * Creatinine within institutional norms for age (i.e. ≤ 2 mg/dL in adults or according to table below in children <18 years) OR creatinine clearance (as estimated by Cockcroft Gault Equation) ≥ 60 mL/min Age (Years) Maximum Serum Creatinine (mg/dL)

      * 5 Years - Serum Creatinine (mg/dL) = 0.8; 5 < age ≤ 10 Years - Serum Creatinine (mg/dL) = 1.0; >10-18 years - Serum Creatinine (mg/dL) = 1.2; > 18 years - Serum Creatinine (mg/dL) = 2.0
    * Serum (alanine aminotransferase/aspartate aminotransferase(ALT/AST)≤ 10x upper limit of normal (ULN) (unless elevated ALT/AST is associated with leukemia involvement of the liver, in which case this criterion will be waived and not disqualify a patient).
    * Total bilirubin ≤ 1.5 mg/dl, except in subjects with Gilbert's syndrome.
    * Cardiac ejection fraction ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an ECHO,
    * No clinically significant ECG findings
    * No clinically significant pleural effusion
    * Baseline oxygen saturation > 92% on room air * if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy); A subject will not be excluded because of pancytopenia ≥ Grade 3 if it is due to disease, based on the results of bone marrow studies.
11. CNS Status Subjects with CNS involvement are eligible as long as there are no overt signs or symptoms that in the evaluation of the investigator would mask or interfere with the neurological assessment of toxicity.
12. Pregnancy Test Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
13. Contraception Subjects of child bearing or child fathering potential must be willing to practice birth control from the time of enrollment on this study and for four (4) months after receiving the preparative regimen or for as long as CD19/CD22-CAR T cells are detectable in peripheral blood.
14. Ability to give informed consent. All subjects ≥ 18 years of age must be able to give informed consent. For subjects <18 years old their legal authorized representative (LAR) (i.e. parent or guardian) must give informed consent. Pediatric subjects will be included in age appropriate discussion and verbal assent will be obtained for those > 7 years of age, when appropriate. If a minor becomes of age during participation of this study, he/she will be asked to reconsent as an adult

EXCLUSION CRITERIA:

1. Recurrent or refractory ALL limited to isolated testicular disease.
2. Hyperleukocytosis (≥ 50,000 blasts/μL) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy
3. History of malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years
4. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
5. Ongoing infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti HCV positive) as the immunosuppression contained in this study will pose unacceptable risk. A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing.
6. CNS disorder such as cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement hat in the judgment of the investigator may impair the ability to evaluate neurotoxicity.
7. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
8. Any medical condition that in the judgement of the sponsor investigator is likely to interfere with assessment of safety or efficacy of study treatment
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
10. Women of child bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
11. In the investigators judgment, the subject is unlikely to complete all protocol required study visits or procedures, including follow up visits, or comply with the study requirements for participation
12. Has primary immunodeficiency or history of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2036-09-10 (Estimated)

PRIMARY OUTCOMES:
Rate of successful manufacture of CD22 CAR T cells | 7-11 days after apheresis
  The percentage of apheresis samples (fresh or frozen) that are successfully processed and expanded to manufacture CD22 CAR T cells that satisfy the target dose level and meet release specifications will be determined for each disease group (ALL or lymphoma).
Safe dose of CD22-CAR T cells in subjects with R/R B-cell malignancies | 28 days after infusion
  Incidence and severity of dose limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD22 CAR T cells, as recorded and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, at target dose of 1 x 10^6 transduced T cells/kg (± 20%).

SECONDARY OUTCOMES:
Clinical activity of CD22-CAR T cells in children and young adults with R/R CD22-expressing B-cell ALL and R/R lymphoma | 28 days after infusion of CD22-CAR T cells
  Clinical activity will be assessed by modified International Working Group response criteria for acute lymphoblastic leukemia (ALL). Results will be reported as best response (i.e. complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PR)) at Day 28 for adult subjects with ALL treated at the target dose.
Clinical activity of CD22-CAR T cells in adults with R/R lymphoma | 3 months after infusion of CD22-CAR T cells
  Clinical activity will be assessed by Lugano response criteria for lymphoma. Results will be reported as best response (i.e. complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PR)) at Month 3 for adult lymphoma/DLBCL subjects treated at Maximum tolerated dose (MTD) /recommended phase 2 dose (RP2D).

CONTACTS AND LOCATIONS:
Overall Officials: Liora Schultz, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No